CLINICAL TRIAL: NCT06415006
Title: Can Shock Indices Be Prognostic Indicators in Sepsis/Septic Shock?
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi (Other)
Responsible Party: Principal Investigator, Furkan Tontu, Doctor of Anesthesiology and Reanimation, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2023-24-20
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Shock, Septic; Hemodynamic Instability
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Sepsis: The group consists of 1,522 patients treated in the intensive care unit for sepsis/septic shock.
  Interventions: Procedure: Measurement of hemodynamic parameters.

INTERVENTIONS:
Procedure: Measurement of hemodynamic parameters. — The measurement and recording of Heart Rate (HR), Systolic Arterial Blood Pressure (ABPsys), Diastolic Arterial Blood Pressure (ABPdias), Mean Arterial Blood Pressure (ABPmean), and age parameters.

SUMMARY:
We evaluated the ability of shock indices and hemodynamic parameters to predict 28-day ICU mortality.

DETAILED DESCRIPTION:
Shock indices and hemodynamic parameters are significant determinants of mortality in adult ICU patients. This study aimed to evaluate the potential of four known shock indices Shock Index (SI), Age-adjusted Shock Index (aSI), Diastolic Shock Index (dSI), and hemodynamic parameters including Heart Rate (HR), Systolic Arterial Blood Pressure (ABPsys), Diastolic Arterial Blood Pressure (ABPdias), and Mean Arterial Blood Pressure (ABPmean) in predicting 28-day ICU mortality in patients diagnosed with sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a preliminary diagnosis of sepsis/septic shock in the intensive care unit
2. Adult patients aged between 18 and 80 years

Exclusion Criteria:

1. Patients under 18 years old
2. Pregnant patients
3. Patients suspected of having COVID-19 pneumonia
4. Patients with incomplete data
5. Patients for whom outcome information is unavailable due to referral to an external center
6. Patients with confirmed COVID-19, validated by thoracic computed tomography images and nasal swab PCR results
7. Patients discharged from the intensive care unit within 24 hours

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: "1,522 patients treated for sepsis/septic shock in the Anesthesiology and Reanimation intensive care unit at Bakırköy Dr. Sadi Konuk Training and Research Hospital."
Sampling Method: Probability Sample
Enrollment: 1522 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Shock Index (SI) | During the first 7 hours in the ICU
  The predictive power of the Shock Index (SI) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
Age-adjusted Shock Index (aSI) | During the first 7 hours in the ICU
  The predictive power of the Age-adjusted Shock Index (aSI) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
Diastolic Shock Index (dSI) | During the first 7 hours in the ICU
  The predictive power of the Diastolic Shock Index (dSI) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
modified Shock Index (mSI) | During the first 7 hours in the ICU
  The predictive power of the modified Shock Index (mSI) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.

SECONDARY OUTCOMES:
Heart Rate (HR) | During the first 7 hours in the ICU
  The predictive power of the Heart Rate (HR) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
Systolic Arterial Blood Pressure (ABPsys) | During the first 7 hours in the ICU
  The predictive power of the Systolic Arterial Blood Pressure (ABPsys) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
Diastolic Arterial Blood Pressure (ABPdias) | During the first 7 hours in the ICU
  The predictive power of the Diastolic Arterial Blood Pressure (ABPdias) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
Mean Arterial Blood Pressure (ABPmean) | During the first 7 hours in the ICU
  The predictive power of the Mean Arterial Blood Pressure (ABPmean) parameter for 28-day mortality in sepsis patients treated in the intensive care unit.
Age | During the first 7 hours in the ICU
  The predictive power of the age for 28-day mortality in sepsis patients treated in the intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Result] Sadeh R, Shashar S, Shaer E, Slutsky T, Sagy I, Novack V, Zeldetz V. Modified Shock Index as a Predictor for Mortality and Hospitalization Among Patients With Dementia. J Emerg Med. 2022 May;62(5):590-599. doi: 10.1016/j.jemermed.2021.12.023. Epub 2022 Feb 16. PMID 35181187
- [Result] Bondariyan N, Vakhshoori M, Sadeghpour N, Shafie D. Prognostic Value of Shock Index, Modified Shock Index, and Age-Adjusted Derivatives in Prediction of In-Hospital Mortality in Patients with Acute Decompensated Heart Failure: Persian Registry of Cardiovascular Disease/ Heart Failure Study. Anatol J Cardiol. 2022 Mar;26(3):210-217. doi: 10.5152/AnatolJCardiol.2021.671. PMID 35346907
- [Result] Pramudyo M, Marindani V, Achmad C, Putra ICS. Modified Shock Index as Simple Clinical Independent Predictor of In-Hospital Mortality in Acute Coronary Syndrome Patients: A Retrospective Cohort Study. Front Cardiovasc Med. 2022 Jun 9;9:915881. doi: 10.3389/fcvm.2022.915881. eCollection 2022. PMID 35757344
- [Result] Kurt E, Bahadirli S. The Usefulness of Shock Index and Modified Shock Index in Predicting the Outcome of COVID-19 Patients. Disaster Med Public Health Prep. 2022 Aug;16(4):1558-1563. doi: 10.1017/dmp.2021.187. Epub 2021 Jun 8. PMID 34099089
- [Result] Gokcek K, Gokcek A, Demir A, Yildirim B, Acar E, Alatas OD. In-hospital mortality of acute pulmonary embolism: Predictive value of shock index, modified shock index, and age shock index scores. Med Clin (Barc). 2022 Apr 22;158(8):351-355. doi: 10.1016/j.medcli.2021.04.035. Epub 2021 Aug 14. English, Spanish. PMID 34404518
- [Result] Kocaoglu S, Karadas A. Comparison of the Effectiveness of Shock Index, Modified Shock Index, and Age Shock Index in COPD Exacerbations. J Coll Physicians Surg Pak. 2022 Sep;32(9):1187-1190. doi: 10.29271/jcpsp.2022.09.1187. PMID 36089718
- [Result] Vang M, Ostberg M, Steinmetz J, Rasmussen LS. Shock index as a predictor for mortality in trauma patients: a systematic review and meta-analysis. Eur J Trauma Emerg Surg. 2022 Aug;48(4):2559-2566. doi: 10.1007/s00068-022-01932-z. Epub 2022 Mar 8. PMID 35258641
- [Result] Zhang TN, Hao PH, Gao SY, Liu CF, Yang N. Evaluation of SI, MSI and DSI for very early (3-day) mortality in patients with septic shock. Eur J Med Res. 2022 Nov 3;27(1):227. doi: 10.1186/s40001-022-00857-y. PMID 36329534
- [Result] Althunayyan SM, Alsofayan YM, Khan AA. Shock index and modified shock index as triage screening tools for sepsis. J Infect Public Health. 2019 Nov-Dec;12(6):822-826. doi: 10.1016/j.jiph.2019.05.002. Epub 2019 May 18. PMID 31113741
- [Result] Georgette N, Michelson K, Monuteaux M, Eisenberg M. A Temperature- and Age-Adjusted Shock Index for Emergency Department Identification of Pediatric Sepsis. Ann Emerg Med. 2023 Oct;82(4):494-502. doi: 10.1016/j.annemergmed.2023.03.026. Epub 2023 May 12. PMID 37178098
- [Result] Gupta S, Alam A. Shock Index-A Useful Noninvasive Marker Associated With Age-Specific Early Mortality in Children With Severe Sepsis and Septic Shock: Age-Specific Shock Index Cut-Offs. J Intensive Care Med. 2020 Oct;35(10):984-991. doi: 10.1177/0885066618802779. Epub 2018 Oct 2. PMID 30278814
- [Result] Avci M, Doganay F. Prognostic Performance of Shock Index, Diastolic Shock Index, Age Shock Index, and Modified Shock Index in COVID-19 Pneumonia. Disaster Med Public Health Prep. 2022 May 2;17:e189. doi: 10.1017/dmp.2022.110. PMID 35492010